CLINICAL TRIAL: NCT02381054
Title: Translation, Cross-Cultural Adaptation and Validation of the US National Cancer Institute's Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) for Italian-speaking Cancer Patients
Brief Title: Translation, Cross-cultural Adaptation and Validation of PRO-CTCAE for Italian-speaking Cancer Patients
Acronym: PRO-CTCAE
Status: Completed | Type: Observational
Sponsor: Italian PRO-CTCAE Study Group (Other)
Collaborators: National Cancer Institute, Naples (Other); F.A.V.O. Italian Federation of Volunteer-Based Cancer Organizations (Unknown); SmithKline Foundation (Unknown); Parma University Hospital (Other); IRCCS AOU San Martino -IST Genoa (Unknown); Istituti Ospitalieri di Cremona (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: Italian PRO-CTCAE
Record Dates: First submitted 2015-02-27; First posted 2015-03-06 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Cancer
Keywords: Patient reported outcomes
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Translation and cross-cultural adaptation phase: In this phase 96 Italian-speaking patients who are receiving cancer treatment or who have completed treatment for cancer within the past six months at one of the participating sites will first be asked to independently complete a series of PRO-CTCAE symptom items in a Patient Questionnaire. Following completion by the participant of the Patient Questionnaire containing PRO-CTCAE items, the interviewer will elicit participants' feedback regarding item comprehension, symptomatic adverse event terms, attribute terms, 7-day recall period, and response options, via a semi-scripted cognitive debriefing interview developed to assure consistency across interviews.
- Test-retest phase: In this phase a minimum of 59 Italian-speaking patients who are receiving cancer treatment will be asked to independently complete the Italian version PRO-CTCAE questionnaire on 2 consecutive business days.

SUMMARY:
The purpose of this study is to see if the Italian language version of a questionnaire about symptoms that patients may have during cancer treatment is understandable to Italian speaking patients. The questionnaire is called the PRO-CTCAE, and was originally developed at the U.S. National Cancer Institute to help get information about patients' symptoms directly from the patients themselves. The Italian version of the questionnaire will be used in future studies to gain a better understanding of patient symptoms.

DETAILED DESCRIPTION:
This study will be conducted in two steps. The first is the Italian translation and cross cultural adaptation of the original US NCI's version of the PRO-CTCAE questionnaire. The questionnaire will be translated and administered to a sample of 96 Italian patients. After protocol amendment in November 2016, the second step was modified and consists of test-retest reliability assessment of the Italian language version of the PRO-CTCAE questionnaire that was developed in the first step, with a minimum of 59 Italian speaking patients to be enrolled. A validation study is planned and will be the subject of a separate protocol.

ELIGIBILITY:
Eligibility Criteria for cross-cultural adaption phase:

Inclusion criteria:

* patients receiving (or who have received within 6 months) chemotherapy or radiotherapy with curative or palliative intent for an advanced cancer at one of the study sites
* ≥18 years of age
* able to speak and understand Italian
* providing written informed consent

Exclusion criteria:

• Patients judged unable to report on their symptoms from the last seven days due to cognitive impairment.

Eligibility Criteria for Validation phase:

Inclusion Criteria:

* ≥18 years of age.
* Patient is able to complete PRO-CTCAE on two consecutive days.
* Patient is actively receivingmedical treatment for cancer or has completed treatment not more than 4 weeks before Visit 1
* Any type of cancer
* Able to complete questionnaire by themselves or with assistance.
* Providing informed written consent.
* Able to speak and understand Italian

Exclusion Criteria:

* Clinically significant cognitive or memory impairment in the opinion of clinical or research staff.
* Other important acute medical conditions that, in the opinion of the Investigator, may prevent compliance..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving or having recently received cancer therapy (chemotherapy, biologic therapy, and or radiation therapy) will be recruited from 17 Italian Cancer Institutes and Hospitals throughout Italy. Sampling will be performed to ensure that the target population is matched for gender, age and area of residence (North, center, and Southern Italy). Recruitment of at least 25% of patients with lower levels of educational attainment (i.e., primary school or no education) will also be ensured.
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-06-22 (Actual)

PRIMARY OUTCOMES:
cultural and linguistic validity of Italian language version of the PRO-CTCAE | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Perrone, Principal Investigator — National Cancer Institute, Naples; Caterina Caminiti, Principal Investigator — Parma University Hospital; Michela Bagnalasta, Principal Investigator — Smith Kline Foundation; Fabio Arpinelli, Principal Investigator — Smith Kline Foundation; Maurizio Bassi, Principal Investigator — Smith Kline Foundation; Pierpaolo Betteto, Principal Investigator — F.A.V.O. Italian Federation of Volunteer-Based Cancer Organizations; Lucia Del Mastro, Principal Investigator — IRCCS AOU San Martino -IST, National Cancer Research Institute; Davide De Persis, Principal Investigator — F.A.V.O. Italian Federation of Volunteer-Based Cancer Organizations; Elisabetta Iannelli, Principal Investigator — F.A.V.O. Italian Federation of Volunteer-Based Cancer Organizations; Anna Lisa Nicelli, Principal Investigator — Smith Kline Foundation; Rodolfo Passalacqua, Principal Investigator — Istituti Ospitalieri Cremona; Camillo Porta, Principal Investigator — Fondazione I.R.C.C.S. Policlinico San Matteo; Jane Bryce, Principal Investigator — National Cancer Institute, Naples
Locations (16):
- Italy (16):
  - IRCCS Istituto Oncologico"Giovanni Paolo II", Bari
  - Ospedale "A.Perrino", Brindisi
  - Istituti Ospitalieri, Cremona
  - IRCCS AOU San Martino -IST, Genova
  - AOU Policlinico G.Martino, Messina
  - Istituto Nazionale Tumori, Milan
  - Istituto Nazionale Tumori - Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto, Padua
  - IRCCS Policlinico S.Matteo, Pavia
  - A.O. Sant'Andrea, Roma
  - Ospedale San Camillo Forlanini, Roma
  - Policlinico Umberto I, Roma
  - Ospedale Civile SS.Annunziata, Sassari
  - Ospedale Valdelsa di Poggibonsi, Siena
  - AOU San Luigi Orbassano, Torino
  - Policlinico Universitario G.B.Rossi, Verona